CLINICAL TRIAL: NCT04991740
Title: A Phase 1 Study of JNJ-78306358, a T Cell Redirecting Bispecific Antibody Targeting HLA-G for Advanced Stage Solid Tumors
Brief Title: A Study of JNJ-78306358 in Participants With Advanced Stage Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109028; 2021-001646-35 (EudraCT Number); 78306358STM1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-08-02; First posted 2021-08-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms
Keywords: Kidney cancer; Ovarian cancer; Colorectal cancer
MeSH Terms: conditions — Neoplasms; Kidney Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with renal cell carcinoma (RCC), ovarian cancer, colorectal cancer (CRC), and other tumor types with sponsor approval will receive JNJ-78306358. The dose will be escalated sequentially based on the decisions of the study evaluation team until the recommended phase 2 dose (RP2D) regimen(s) have been identified.
  Interventions: Drug: JNJ-78306358
- Part 2: Dose Expansion (Experimental): Participants with RCC, ovarian cancer, CRC and other types of tumors will receive JNJ-78306358 at the RP2D regimen(s) determined in Part 1.
  Interventions: Drug: JNJ-78306358

INTERVENTIONS:
Drug: JNJ-78306358 — JNJ-78306358 will be administered.

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose (RP2D) regimen(s) of JNJ-78306358 in Part 1 (Dose Escalation) and to determine the safety of JNJ-78306358 at the RP2D regimen(s) in Part 2 (Dose Expansion).

DETAILED DESCRIPTION:
JNJ-78306358 is a bispecific antibody binding to CD3 on T cells and human leukocyte antigen G (HLA-G) on cancer cells. The study consists of a screening phase, a treatment phase, and a post-treatment follow-up phase. Study evaluations include safety, pharmacokinetics, biomarkers, immunogenicity, and efficacy (disease evaluations). The total study duration will be up to 2 years 4 months.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed, metastatic or unresectable solid tumor of one of the following types:

  a. Renal Cell Carcinoma (RCC): clear cell or papillary carcinoma, b. ovarian cancer: high grade serous epithelial ovarian; primary peritoneal or fallopian tube cancer; 1. low grade or non-serous histologies are not allowed; c. colorectal cancer (CRC); d. other tumor types (including lung adenocarcinoma, endometrial cancer, and pancreas cancer) may be enrolled with sponsor approval
* Measurable or evaluable disease: a. Part 1: either measurable or evaluable disease; b. Part 2: at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Participants with ovarian cancer without a measurable lesion must have disease evaluable per RECIST version1.1 (example ascites) or have Cancer antigen 125 (CA 125) greater than (>) 2*upper limit of normal (ULN) within 2 weeks prior to first dose of study drug
* Progressed during or after the following prior therapies for metastatic disease, unless participant was ineligible to receive them: a) RCC: clear cell histology: an antiangiogenic agent and an immune checkpoint inhibitor, administered as 1 or more lines of therapy. For papillary renal carcinoma 1 line of systemic therapy; b. CRC: at least 2 lines of therapy including a fluoropyrimidine, oxaliplatin, and irinotecan given with or without antiangiogenic therapies or epidermal growth factor receptor (EGFR) antibodies. In addition, prior treatment with anti-programmed cell death protein 1 (PD1) antibody is required for high microsatellite instability (MSI-H) CRC; c. ovarian cancer: at least 2 lines of therapy, including at least 1 line with platinum. Maintenance therapy after completion of platinum-containing regimen, example with bevacizumab or a poly- Adenosine di-phosphate (ADP) ribose polymerase inhibitor will not count as a separate line of therapy; d. other tumor types: at least 2 lines of systemic therapy
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Selected participants in pharmacokinetics/pharmacodynamic (PK/PD) cohorts and in Part 2 must agree to undergo the mandatory tumor biopsies

Exclusion Criteria:

* Active central nervous system involvement
* Toxicity from prior anticancer therapy has not resolved to baseline levels or to Grade less than or equal to (<=) 1 (except alopecia, vitiligo, peripheral neuropathy, or endocrinopathies that are stable on hormone replacement, which may be Grade 2)
* Clinically significant pulmonary compromise
* Autoimmune or inflammatory disease requiring systemic steroids or other immunosuppressive agents (example, methotrexate or tacrolimus) within 1 year prior to first dose of study drug
* Solid organ or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-10-24 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Incidence of Adverse Events (AEs) | Up to 2 years and 4 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 2 years and 4 months
  Number of participants with AEs by severity will be reported. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) events, which will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 21 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of JNJ-78306358 | Up to 2 years and 4 months
  Cmax is defined as maximum serum concentration of JNJ-78306358.
Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-78306358 | Up to 2 years and 4 months
  Tmax is defined as time to reach maximum observed serum concentration of JNJ-78306358.
Area Under the Serum Concentration-time Curve From Time t1 to t2 (AUC[t1-t2]) of JNJ-78306358 | Up to 2 years and 4 months
  AUC(t1-t2) is defined as the area under the serum concentration-time curve from time t1 to t2.
Accumulation Ratio (RA) of JNJ-78306358 | Up to 2 years and 4 months
  RA is calculated as area under the plasma concentration-time curve from time zero to 24 hours (AUC [0-24]) value at steady state divided by AUC (0-24) value after first dose.
Number of Participants with Anti-JNJ-78306358 Antibodies | Up to 2 years and 4 months
  Number of participants with anti-JNJ-78306358 antibodies will be reported.
Overall Response Rate (ORR) | Up to 2 years and 4 months
  ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR), according to response evaluation criteria in solid tumors (RECIST) version 1.1 and gynecological cancer inter group (GCIG) Cancer antigen 125 (CA 125) response criteria (for ovarian cancer participants only).
Duration of Response (DOR) | Up to 2 years and 4 months
  Duration of response (DOR) will be calculated among responders (PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the RECIST version 1.1 response criteria and GCIG CA 125 response criteria (for ovarian cancer participants only) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Israel (2):
  - Rambam Medical Center, Haifa
  - Sourasky Medical Center, Tel Aviv
- Spain (3):
  - Hosp. Univ. Vall D Hebron, Barcelona
  - Hosp. Univ. Fund. Jimenez Diaz, Madrid
  - Hosp. Univ. Hm Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Geva R, Vieito M, Ramon J, Perets R, Pedregal M, Corral E, Doger B, Calvo E, Bardina J, Garralda E, Brown RJ, Greger JG, Wu S, Steinbach D, Yao TS, Cao Y, Lauring J, Chaudhary R, Patel J, Patel B, Moreno V. Safety and clinical activity of JNJ-78306358, a human leukocyte antigen-G (HLA-G) x CD3 bispecific antibody, for the treatment of advanced stage solid tumors. Cancer Immunol Immunother. 2024 Aug 6;73(10):205. doi: 10.1007/s00262-024-03790-7. PMID 39105878